CLINICAL TRIAL: NCT02570048
Title: Tinnitus Alleviation Via Sensory Substitution (Modulation of Tinnitus Through Simultaneous Auditory and Transcutaneous Tactile Stimulation of the Tongue).
Brief Title: 1 Tinnitus Alleviation Via Sensory Substitution
Status: Completed | Type: Observational
Sponsor: MuteButton (Industry)
Responsible Party: Sponsor
Other Study IDs: Tinnitus pilotV1
Record Dates: First submitted 2015-09-28; First posted 2015-10-07 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Experimental: Mutebutton intervention: This one armed trail will recruit participants who have been diagnosed with Tinnitus for a minimum of 6 months. Participants will use the Mutebutton device in their own home for 30 minutes every day for 12 weeks. The intervention requires sitting in a quiet space with the earphones on and the tongue tip placed on their tongue.
  Interventions: Device: Mutebutton intervention

INTERVENTIONS:
Device: Mutebutton intervention — Participants are asked to use the MuteButton daily for 30-40 minutes.They receive 'pink noise' through headphones and transcutaneous stimulation on the tongue using a 'lollypop' sensor that sits on the anterior section (tip) of the tongue.

SUMMARY:
This is a novel experimental device 'MuteButton' can affect the awareness of tinnitus. Sound that arrives at the ears naturally will be presented in the form of touch patterns on the tongue. By learning to associate the sounds in the ears with the sound patterns on the tongue, investigators aim to demonstrate that the brain will learn to discriminate the real sounds from legitimate external sounds from the imaginary tinnitus sounds that are created inside the brain. Tinnitus is an audiological condition most commonly described as 'ringing in the ears' that affects an estimated 40 million people globally (American Tinnitus Association; Royal National Institute for Deaf). More accurately, tinnitus is the perception of illusory sound that has no legitimate external source and normally arises from a small number of underlying neuropathologies. There are broadly two categories of tinnitus Somatic Tinnitus and Hearing Loss Related Tinnitus.

MuteButton is indicated for the treatment of permanent intractable subjective tinnitus. The study is intended to show the efficacy of MuteButton treatment in alleviating tinnitus. The objective of the study will be to determine the impact of acoustic and tactile multi-modal neuromodulation on symptoms of permanent intractable tinnitus as measured by objective and subjective measures including Minimum Masking Level (MML), Tinnitus Loudness Masking (Tinnitus Loudness Masking), Tinnitus Handicap Inventory (THI) and Visual Analogue Scale (VAS).

DETAILED DESCRIPTION:
This study will be a prospective single arm pilot study. It will be conducted with approval from the Research Ethics Committee of NUI Maynooth and The Hermitage Medical Clinic Lucan in collaboration with Mutebutton Ltd, Nova UCD. This study will be conducted over a 16-week period with 60 suffering from permanent intractable tinnitus (>6 months) and with an accompanying/ co-existing high-frequency hearing-loss. Participants will be screened for a 4-week run-in period prior to commencement of treatment where baseline measures will be obtained and sampled every 2 weeks. Following this run-in period they will receive treatment for 10 weeks and will be followed up 2 weeks post-treatment. For the duration of the study they will be assessed every 2 weeks in the clinical environment. Participants will be given the IFU (Appendix 3) along with the device and given step by step instructions on how to use it, and a detailed description of each control, indicator and connection. Participants will use the MuteButton device for minimum of 1 hour a day for a period of 10 weeks.

The efficacy of the intervention will be assessed by the change in several psychoascoutic assessments assessed every at each of the 6 follow up visits with the investigators at 2 week intervals.

The Psychoacoustic Assessment will include:

Tinnitus Matching (Pitch) - symptom severity Tinnitus Loudness Matching (TLM ) - symptom severity Minimum Masking Level (MML) - symptom severity

Questionnaires to be utilised will include:

Visual Analogue Scale (VAS) - symptom severity Tinnitus Handicap Inventory (THI) - symptom severity A primary endpoint at 16 weeks is to show a reduction in a THI, and psychoacoustic assessment will be established. Secondary endpoint will include reduction in MML, and psychoacoustic assessment will be established.

ELIGIBILITY:
Inclusion Criteria:

* aged <65 years
* suffering from subjective intractable tinnitus
* tinnitus > 6 months
* tinnitus associated with an age or noise related sensory-neural hearing loss
* have sound English reading, comprehension and written skills
* Able and willing to participate in the study for the 16 weeks duration.
* Informed consent

Exclusion Criteria:

* Ulceration of oral cavity or tongue, oral mucosa or significant intra oral disease - to mitigate risk of further aggravation these symptoms
* Meniere's Disease - due to the fluctuating hearing loss patients normally present with
* Hyperacusis - to avoid further aggravation of sensitivity of sound
* Current medical legal cases regarding tinnitus or hearing - in order to avoid any conflict of interest
* Undergoing any treatment for tinnitus - in order to accurately measure the independent effect of the intervention.
* Pacemakers - due to potential magnetic interference.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be persons who are diagnosed as having tinitus by an audiologists that are at least 18 years of age. It is expected that the user age distribution will be skewed towards an older deomographic due to the increased prevalence of hearing loss-related tinnitus in the elderly.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Number of participants who achieve a clinically significant reduction in Tinnitus Handicap Inventory (THI) score | 12 weeks

SECONDARY OUTCOMES:
Difference in mean Visual Analogue Scale (VAS) score from before after intervention | 12 weeks
Difference in mean Tinnitus Loudness Matching (TLM) score before and after intervention. | 12 weeks
Difference in mean Minimum Masking Level (MML) score intervention before and after intervention. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Hamilton, Principal Investigator — MuteButton
Locations (1):
- Hermitage Medical Clinic, Lucan, Dublin, Ireland